CLINICAL TRIAL: NCT02895802
Title: Assessing the Feasibility of the Use of Visual Aids in Patient Education in Adults With Down Syndrome (DS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 6360
Record Dates: First submitted 2016-08-27; First posted 2016-09-12 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2019-01

CONDITIONS: Down Syndrome
Keywords: down syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Verbal instructions with picture diagram (Other): hand washing is scored prior and after educational intervention with verbal instructions of handwashing and a picture diagram of handwashing.
  Interventions: Behavioral: Verbal instructions with picture diagram
- Verbal instructions with video of ADSC (Other): hand washing is scored prior and after educational intervention with verbal instructions of handwashing and a video of the adult down syndrome center
  Interventions: Behavioral: Verbal instructions with video of ADSC
- verbal instructions w. video of w/o DS (Other): hand washing is scored prior and after educational intervention with verbal instructions of handwashing and viewing an educational video depicting a person without down syndrome washing their hands.
  Interventions: Behavioral: verbal instructions w. video of w/o DS
- verbal instructions w.video w/DS (Other): hand washing is scored prior and after educational intervention with verbal instructions of handwashing and watching an educational video depicting a person with down syndrome washing their hands.
  Interventions: Behavioral: verbal instructions w. video w/DS

INTERVENTIONS:
Behavioral: Verbal instructions with picture diagram — verbal instructions and picture diagram
  Arms: Verbal instructions with picture diagram
Behavioral: Verbal instructions with video of ADSC — Verbal instructions and watching video depicting ADSC
  Arms: Verbal instructions with video of ADSC
Behavioral: verbal instructions w. video of w/o DS — verbal instructions and watching video depicting person without DS washing her hands
  Arms: verbal instructions w. video of w/o DS
Behavioral: verbal instructions w. video w/DS — verbal instructions and watching video depicting person with DS washing his hands
  Arms: verbal instructions w.video w/DS

SUMMARY:
Purpose: To assess the feasibility of using videos depicting people with DS to teach other adults with DS to perform healthy behaviors.

Hypothesis: Videos of adults with DS performing healthy behaviors is a more effective way to promote healthy behaviors by adults with DS than other methods tested.

This project will study whether videos showing a person with DS washing his hands correctly can improve hand washing by other adults with DS.

DETAILED DESCRIPTION:
The subjects will be recruited and identified and consented. Subjects will be randomized to one of 4 groups.

i. Verbal instructions on hand washing with pictures (using the Illinois department of public health tools) ii. Verbal instructions on hand washing and video of the ADSC iii. Verbal instructions on hand washing and video of an adult without DS washing his hands iv. Verbal instructions on hand washing and video of an adult with DS washing his hands.

Videos of the handwashing process will be taken pre intervention and then again post intervention.

Scoring assessments will be completed upon review of the 2 files by 2 separate study team members, the second of which will be blinded to the information they will be reviewing.

ELIGIBILITY:
Inclusion Criteria:

* People with Down syndrome receiving care at Advocate
* No known sensitivity to soap

Exclusion Criteria:

* Pregnant women, prisoners
* Known sensitivity to soap

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Score on handwashing checklist | 2 minutes
  2 minute videos will be reviewed and scored twice. First by research coordinator then by blinded reviewer. Scores will be compared and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Chicoine, MD, Principal Investigator — Advocate Health and Hospitals Corporation
Locations (1):
- Adult Down Syndrome Center / Russell Institute for Research and Innovation, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ram G, Chinen J. Infections and immunodeficiency in Down syndrome. Clin Exp Immunol. 2011 Apr;164(1):9-16. doi: 10.1111/j.1365-2249.2011.04335.x. Epub 2011 Feb 24. PMID 21352207
- [Result] Parker RM, Ratzan SC, Lurie N. Health literacy: a policy challenge for advancing high-quality health care. Health Aff (Millwood). 2003 Jul-Aug;22(4):147-53. doi: 10.1377/hlthaff.22.4.147. PMID 12889762
- [Result] Lee RL, Lee PH. To evaluate the effects of a simplified hand washing improvement program in schoolchildren with mild intellectual disability: a pilot study. Res Dev Disabil. 2014 Nov;35(11):3014-25. doi: 10.1016/j.ridd.2014.07.016. Epub 2014 Aug 12. PMID 25124699
- [Result] Kagohara DM, van der Meer L, Ramdoss S, O'Reilly MF, Lancioni GE, Davis TN, Rispoli M, Lang R, Marschik PB, Sutherland D, Green VA, Sigafoos J. Using iPods((R)) and iPads((R)) in teaching programs for individuals with developmental disabilities: a systematic review. Res Dev Disabil. 2013 Jan;34(1):147-56. doi: 10.1016/j.ridd.2012.07.027. Epub 2012 Aug 30. PMID 22940168
- [Result] Global consensus conference: final recommendations. Am J Infect Control. 1999 Dec;27(6):503-13. doi: 10.1016/s0196-6553(99)70029-5. No abstract available. PMID 10586155